CLINICAL TRIAL: NCT01226017
Title: A Possible Effect of Oxytocin During Interaction Between Humans and Animals
Acronym: Oxytocin2010
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Life Sciences (Other)
Responsible Party: Principal Investigator, Gunn Pedersen, MPh, Norwegian University of Life Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010/1589
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Animal Assisted Therapy
Keywords: Oxytocin; Animal Assisted therapy; Farm animals; Healthy nursing students
MeSH Terms: interventions — Blood Specimen Collection; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Measuring oxytocin level in blood — Blood sampling and instruments measuring anxiety and stress
  Other Names: Oxytocin

SUMMARY:
The purpose of this pilot study is to investigate the possible change of Oxytocin level in human blood after positive interaction with farm animals.

DETAILED DESCRIPTION:
The purpose of this pilot study is to investigate the possible change of Oxytocin level in human blood after positive interaction with farm animals and filling in instruments measuring anxiety and stress.

ELIGIBILITY:
Inclusion Criteria:

* woman
* age 20-30 years old
* physical capable of being in a farm environment and have contact with cows

Exclusion Criteria:

* pregnancy
* breastfeeding
* anxiety for blood sampling
* anxiety for animals
* allergies
* psychiatric diagnoses
* medication

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Measuring the possible change in Oxytocin level in human blood during intervention with farm animals. | Start medio October 2010, and end December 2011 (14 months)
  Blood sampling will be drawn at baseline, before intervention starts, and 5 minutes after start. 3rd sample will be drawn 15 minutes after start. Total time of intervention is 15 minutes.

SECONDARY OUTCOMES:
Self evaluation of anxiety and coping strategies. | Start medio October 2010, and end December 2011 (14 months)
  Spielberger State Anxiety Inventory (SSAI) (Spielberger et al, 1979)and Coping Strategies Scale of the Pressure Management Indicator (Williams & Cooper, 1998.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Berget, PhD, Principal Investigator — Norwegian University of Life Sciences
Locations (1):
- Norwegian University of Life sciences, Aas, Aas, Norway